CLINICAL TRIAL: NCT05223335
Title: Clopidogrel Monotherapy in High Bleeding Risk Patients Undergoing Percutaneous Coronary Interventions: A Safety Assessment, Pilot Study to Reduce Post-Discharge Bleeding
Brief Title: Clopidogrel Monotherapy in Patients With High Bleeding Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-011053
Record Dates: First submitted 2022-01-06; First posted 2022-02-03 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Bleeding Complications
Keywords: Antiplatelet medications; Blood thinners; Stent thrombosis; Percutaneous Coronary Intervention
MeSH Terms: interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Genotype-Guided Therapy (Experimental): Subjects with high bleeding risk (HBR) on dual antiplatelet therapy (DAPT) with clopidogrel and aspirin, that have undergone successful percutaneous coronary intervention (PCI) will be stratified by the CYP2C19 loss-of-function (LOF) allele within one week of DAPT initiation. In this group, subjects identified as CYP2C19*2 or*3 LOF allele carrier will be given prasugrel or ticagrelor monotherapy.
  Interventions: Drug: Prasugrel; Drug: Tricagrelor
- Conventional Therapy (Active Comparator): Subjects with high bleeding risk (HBR) on dual antiplatelet therapy (DAPT) with clopidogrel and aspirin, that have undergone successful percutaneous coronary intervention (PCI) will be stratified by the CYP2C19 loss-of-function (LOF) allele within one week of DAPT initiation. In this group, subjects identified as CYp2C19*2 or*3 LOF allele non-carriers will continue with clopidogrel monotherapy.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 75 mg/day
  Arms: Conventional Therapy
Drug: Prasugrel — 60 mg bolus then 10 mg daily
  Arms: Genotype-Guided Therapy
Drug: Tricagrelor — 180 mg bolus then 90 mg twice daily
  Arms: Genotype-Guided Therapy

SUMMARY:
The goal of this research is to show that a shorter duration of two antiplatelet medications (compared to the standard of care) is safe and effective while reducing the risk of bleeding complications. Bleeding complications can cause significant problems (hospitalizations, need for blood transfusions, and even death) for patients on antiplatelet medications after coronary stents. Researchers hope to show that reducing the time on two antiplatelet agents in patients at high risk for these bleeding complications will reduce the number of bleeding events while not causing any increase in cardiovascular complications (heart attack, stent malfunction, death).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent in adults
* Successful percutaneous coronary intervention (PCI) [no non-fatal myocardial infarction (MI)/stroke/repeat target revascularization/bleeding/acute kidney injury].
* Academic research consortium-high bleeding risk (ARC-HBR) score ≥ 4.

Exclusion Criteria:

* Chronic use of warfarin or direct oral anticoagulant (DOAC).
* Unsuccessful PCI (see above).
* Lesions with angiographic thrombus.
* Prior PCI within 6 months.
* Planned PCI or surgical intervention to treat any cardiac or noncardiac condition within 6 months.
* High risk lesion/stent characteristics (> 50% unprotected left main disease, bifurcation disease requiring 2 stents technique, rotational atherectomy.
* Vein graft.
* Unprotected left main intervention or history of definite stent thrombosis.
* Women of child-bearing age unless negative pregnancy test is done.
* Life expectancy < 1 year.
* Known drug/alcohol dependence.
* Assessment that the patient will not be compliant with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Ingraham BS, Huxley SB, Lane CM, Gulati R, Lewis BR, Jaffe AS, Bell MR, Lerman A, Pereira NL, Moyer AM, Baudhuin LM, Rihal CS, Singh M. Genotype-Guided P2Y12 Inhibitor Monotherapy Within 7 Days of Percutaneous Coronary Intervention in High Bleeding Risk Patients: The CHAMP Trial - A Pilot Study and Safety Assessment. Mayo Clin Proc. 2025 Jan;100(1):94-108. doi: 10.1016/j.mayocp.2024.05.030. Epub 2024 Nov 26. PMID 39601743
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Genotype-Guided Therapy: Subjects with high bleeding risk (HBR) on dual antiplatelet therapy (DAPT) with clopidogrel and aspirin, that underwent successful percutaneous coronary intervention (PCI) were stratified by the CYP2C19 loss-of-function (LOF) allele within one week of DAPT initiation. In this group, subjects identified as CYP2C19*2 or*3 LOF allele carrier were given prasugrel or ticagrelor monotherapy.
  Prasugrel: 60 mg bolus then 10 mg daily
  Tricagrelor: 180 mg bolus then 90 mg twice daily
- Conventional Therapy: Subjects with high bleeding risk (HBR) on dual antiplatelet therapy (DAPT) with clopidogrel and aspirin, that underwent successful percutaneous coronary intervention (PCI) were stratified by the CYP2C19 loss-of-function (LOF) allele within one week of DAPT initiation. In this group, subjects identified as CYp2C19*2 or*3 LOF allele non-carriers continued with clopidogrel monotherapy.
  Clopidogrel: 75 mg/day
Period: Overall Study
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Started | 29 | 69
Completed | 29 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype-Guided Therapy | Conventional Therapy | Total
Number analyzed (Participants) | 29 | 69 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (11.7) | 75.3 (10.8) | 74.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 23 | 34
  Male | 18 | 46 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 69 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 26 | 68 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 69 | 98

OUTCOME MEASURES:

1. Primary Outcome: Ischemic Risk Post-PCI in High Bleed Risk Patients With Genotype-guided Single Antiplatelet Therapy
Description: The number of participants to experience ischemic events as defined as cardiac deaths, spontaneous myocardial infarctions (MIs) and stent thrombosis after percutaneous intervention (PCI).
Time Frame: Through study completion, approximately 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Number analyzed (Participants) | 29 | 69
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 90 days
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/69
Other Adverse Events (participants affected / at risk) | 0/29 | 3/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype-Guided Therapy (N=29) | Conventional Therapy (N=69)
Possible Stent Thrombosis (Vascular disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype-Guided Therapy (N=29) | Conventional Therapy (N=69)
BARC 3 bleeding event (Vascular disorders) | 0 | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05223335/Prot_SAP_001.pdf